CLINICAL TRIAL: NCT06060600
Title: A Retrospective Analysis of Suramin Treatment for Stage 1 Trypanosoma Brucei Rhodesiense Human African Trypanosomiasis (S1 TBR HAT) in Uganda and Malawi
Brief Title: A Retrospective Analysis of Suramin Treatment for Stage 1 TBR
Status: Completed | Type: Observational
Sponsor: Paxmedica (Industry)
Responsible Party: Sponsor
Other Study IDs: PAX-HAT-301
Record Dates: First submitted 2023-09-12; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Trypanosoma Brucei Rhodesiense; Infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Natural History Cohort:: * Treatment records from a cohort of approximately 200 patients who were hospitalized between 1901 and 1910 during the 1900-1920 HAT epidemic
  * Treatment records must have sufficient information for analysis including:
    * Demographic data: age or sex must be included
    * Diagnosis: HAT diagnosis is confirmed by blood or lymph gland fluid analysis and parasites observed or HAT symptoms during the epidemic. For example, if the records state that a lymph node biopsy was performed, any result of the biopsy (e.g., documentation that trypanosomes were observed), a documentation of the HAT diagnosis, or mention of HAT symptoms such as sleepiness or excess sleeping are all acceptable. Symptoms alone are not sufficient, but a notation of biopsy and mention of HAT symptoms is acceptable.
    * Outcome: An outcome is required; any mention of a clinical outcome is acceptable.
- Retrospective cohort: The hospital records of TBR HAT patients will be examined for date of symptom onset (if available) and hospital admission, race, sex, age, geographic area of origin, parasites, concomitant medications and illnesses, co-infections, and disease stage. Patients are normally screened for HAT and other tropical diseases using standard parasitological World Health Organization (WHO) criteria. Briefly, blood is obtained from the patients and checked for the presence of trypanosomes using direct wet smear and capillary centrifugation technique methods. Disease stage determination is by examination of CSF using the WHO criteria which classify patients with the presence of trypanosomes in the CSF and/or a WBC count >5 cells/mm3 as Stage 2 TBR HAT. Stage 2 patients would be disqualified from inclusion in the study.

SUMMARY:
The study will include TBR HAT patients treated with suramin between 2000 and 2020 at three sites in Uganda and Malawi A natural history cohort composed of source data from approximately 200 patients from a published epidemiological study will be used as a comparator.

This study's objectives are to evaluate the efficacy and safety of suramin in the Stage 1 treatment of TBR HAT.

DETAILED DESCRIPTION:
The study will include TBR HAT patients treated with suramin between 2000 and 2020 at three sites in Uganda and Malawi (e.g., the retrospective suramin-treated cohort). The study will include all the approximately 145 patients who are deemed eligible through chart review and who have sufficient data. A natural history cohort composed of source data from approximately 200 patients from a published epidemiological study will be used as a comparator.

The primary objective is to determine whether standard of care treatment with suramin, as currently practiced in Uganda and Malawi, leads to better health outcomes in patients with S1 TBR HAT than observed in a natural history cohort with source data from a published epidemiologic study.

ELIGIBILITY:
Inclusion Criteria:

* Suramin-treated cohort:

  * Patient records must meet all the following criteria to be included in the suramin-treated cohort:
  * Male or female of any age; age or sex must be included.
  * Treatment with at least four full doses of suramin (not including the test dose).
  * Onset date or duration of symptoms associated with S1 TBR HAT is available.
  * An outcome is required; any mention of a clinical outcome is acceptable.
  * Must live in an area endemic for TBR HAT
  * Documented HAT diagnosis
  * Positive parasitology for HAT (observed in blood sample or a standard test).

Natural History cohort:

* Treatment records from a cohort of approximately 200 patients who were hospitalized between 1901 and 1910 during the 1900-1920 HAT epidemic
* Treatment records must have sufficient information for analysis including:

  * Demographic data: age or sex must be included
  * Diagnosis: HAT diagnosis is confirmed by blood or lymph gland fluid analysis and parasites observed or HAT symptoms during the epidemic. For example, if the records state that a lymph node biopsy was performed, any result of the biopsy (e.g., documentation that trypanosomes were observed), a documentation of the HAT diagnosis, or mention of HAT symptoms such as sleepiness or excess sleeping are all acceptable. Symptoms alone are not sufficient, but a notation of biopsy and mention of HAT symptoms is acceptable.
  * Outcome: An outcome is required; any mention of a clinical outcome is acceptable.

Exclusion Criteria:

Patient records that meet any of the following criteria will be excluded from the suramin-treated cohort:

* Reported duration of symptoms for more than 2 months at time of presentation at a healthcare facility.
* Stage 2 TBR HAT as determined by examination of cerebrospinal fluid (CSF) using WHO criteria, which classify patients with the presence of trypanosomes in the CSF and/or a WBC count >5 cells/mm3 as Stage 2 TBR HAT at time of presentation to a healthcare facility.
* Evidence of Stage 2 TBR HAT symptoms at time of presentation to a healthcare facility.
* Required medication treatment for Stage 2 illness (melarsoprol) prior to time of presentation to a healthcare facility.
* Known to have had Trypanosoma Brucei Gambiense (TBG) HAT or became ill while travelling from an area known to be endemic for TBG HAT
* Duration of HAT symptoms for more than 6 months. Survival for more than 6 months with TBR HAT is unlikely.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patient charts will be retrieved from three major TBR HAT treatment centers. The study will include approximately 145 patients with S1TBR HAT who have sufficient clinical data for analysis. The study will also include a natural history cohort of the eligible subset of the approximately 200 patients from the 1900-1920 TBR HAT epidemic who were hospitalized in the years 1901 through 1910; some of these patients received experimental treatments such as arsenic which may have had some temporary clinical improvement, but none received any treatment with demonstrated efficacy.
Sampling Method: Non-Probability Sample
Enrollment: 345 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-08-02 (Actual); Study Completion 2023-08-02 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint is survival of patients treated with suramin compared to the natural history cohort. | 30 Days
  The primary efficacy analysis will compare the proportion alive and not meeting any of the following criteria
  * Death (both cohorts).
  * Progression from Stage 1 to Stage 2 TBR HAT as defined by meeting any of the following:
    * presence of TBR trypanosomes in the cerebrospinal fluid (CSF)
    * abnormal symptoms .
    * presence of TBR HAT symptoms for more than 2 months
    * Use of melarsoprol for clinical worsening or treatment failure
  * Moribund status

SECONDARY OUTCOMES:
The secondary objective is to describe the safety and tolerability of suramin. | 30 Days
  • Incidence of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: jennifer L bonfrisco, Study Director — Paxmedica
Locations (1):
- PaxMedica, Tarrytown, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided